CLINICAL TRIAL: NCT04389762
Title: Lactobacillus Plantarum PS128 May Improve Off Duration in Parkinson's Disease: a Pilot Study
Brief Title: PS128 May Improve Off Duration on Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Lu Neurological Clinic (Other)
Responsible Party: Principal Investigator, CHIN-SONG LU, Professor, Professor Lu Neurological Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS128-02
Record Dates: First submitted 2020-04-30; First posted 2020-05-15 (Actual); Results first posted 2025-06-25 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PS128 (Experimental): daily ingestion of Lactobacillus plantarum PS128 capsules
  Interventions: Dietary Supplement: daily ingestion of Lactobacillus plantarum PS128

INTERVENTIONS:
Dietary Supplement: daily ingestion of Lactobacillus plantarum PS128 — daily ingestion of 60 billion colony forming unit (CFU) of Lactobacillus plantarum PS128 (30 billion CFU/capsule)

SUMMARY:
The purpose of this study is to investigate the short term effects (12 Weeks) of Lactobacillus plantarum PS128 (PS128) on Parkinson's disease (PD) symptoms.

DETAILED DESCRIPTION:
This study is designed to examine the extent to which L. plantarum PS128 can improve symptoms in PD patients. L. plantarum PS128 is a psychobiotic that regulates the level of dopamine in specific brain regions. Patients with PD will receive PS128 treatment for 12 weeks. Symptoms of PD will be clinically evaluated before and after the treatment, and the results will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with idiopathic Parkinson's Disease
* According to the record of ON / OFF diary for 3 consecutive days, the patient's daily off periods must be more than 3 hours a day.
* Between ages of 40-80 years old.

Exclusion Criteria:

* Patients on antibiotics within the preceding one month
* Patients using of other probiotic products (sachet, capsule or tablet) within the preceding two weeks
* Have undergone surgery of liver, bladder, or gastrointestinal tract
* Have current or history of inflammatory bowel disease
* Have history of cancer
* Known allergy to probiotics
* Patients with comorbid dementia (Mini-Mental State Examination score ≤ 26) or major depression (The Beck Depression Inventory-II score ≥ 29)
* Have received deep brain stimulation
* Patients receiving artificial enteral or intravenous nutrition

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2020-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Song Lu, MD, Principal Investigator — Professor Lu Neurological Clinic
Locations (1):
- Professor Lu Neurological Clinic, Taoyuan, Guishan Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu CS, Chang HC, Weng YH, Chen CC, Kuo YS, Tsai YC. The Add-On Effect of Lactobacillus plantarum PS128 in Patients With Parkinson's Disease: A Pilot Study. Front Nutr. 2021 Jun 30;8:650053. doi: 10.3389/fnut.2021.650053. eCollection 2021. PMID 34277679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants aged between 40 to 80 who were diagnosed with idiopathic Parkinson's Disease with daily off periods more than 3 hours were enrolled from June 2019 to June 2020. All the participants were administered two capsules containing PS128 (30 billion colony-forming units per capsule) daily for 12 weeks.
Period: Overall Study
Arm/Group | PS128
Started | 26
Completed | 25
Not Completed | 1

BASELINE CHARACTERISTICS:
Population: Parkinson's disease patients between ages of 40-80 years old, according to the record of ON / OFF diary for 3 consecutive days, the patient's daily off periods must be more than 3 hours a day.
Arm/Group | PS128
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 25
Age at onset [Mean (Standard Deviation); unit: years] | 51.72 (6.59)

OUTCOME MEASURES:

1. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale (UPDRS)
Description: The UPDRS scores is a rating tool used to gauge the course of Parkinson's disease in patients. The minimum total score possible is 0 and the maximum total score possible is 199. Higher values represent a worse outcome.
Time Frame: Baseline to Week 12 assessed on medication
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PS128
Number analyzed (Participants) | 25
score on a scale
  pre | 33.00 (10.65)
  post | 29.24 (10.26)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.003, t-test, 2 sided

2. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale Part III (UPDRSIII) "OFF" Period
Description: The UPDRS III scores is subscores of UPDRS, it indicates motor function of PD symptoms. The minimum possible total score is 0 and the maximum possible total score is 108. Higher values represent a worse outcome.
Time Frame: Baseline to Week 12 assessed off medications
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PS128
Number analyzed (Participants) | 25
score on a scale
  pre | 27.16 (7.11)
  post | 24.08 (8.20)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.004, t-test, 2 sided

3. Primary Outcome: Change in Unified Parkinson's Disease Rating Scale Part III (UPDRSIII) "ON" Period
Description: as for outcome 2
Time Frame: Baseline to Week 12 assessed on medications
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PS128
Number analyzed (Participants) | 25
score on a scale
  pre | 17.56 (6.92)
  post | 15.00 (7.76)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.007, t-test, 2 sided

4. Primary Outcome: Change in Patient "ON-OFF" Diary Recording "OFF" Period
Description: "ON-OFF" motor fluctuations are rapid changes in mobility during which PD patients report sudden shifts from adequate mobility to mobility, usually within a few seconds or minutes. The 24-hour diary is divided into 30-minute sections and only mark one answer for each half hour period. It is to know how much time each patient spends in the different Parkinson's states. Higher hours in "OFF" period represent better outcome.
Time Frame: Record for 3 consecutive days prior to Baseline and Week 12 visits by patient-self
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PS128
Number analyzed (Participants) | 25
hours
  pre | 6.52 (1.66)
  post | 5.72 (2.64)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.040, t-test, 2 sided

5. Primary Outcome: Change in Patient "ON-OFF" Diary Recording "ON" Period
Description: Outcome Measure Description: "ON-OFF" motor fluctuations are rapid changes in mobility during which PD patients report sudden shifts from adequate mobility to mobility, usually within a few seconds or minutes. The 24-hour diary is divided into 30-minute sections and only mark one answer for each half hour period. It is to know how much time each patient spends in the different Parkinson's states. Higher hours in "ON" period represent worse outcome.
Time Frame: Record for 3 consecutive days prior to Baseline and Week 12 visits by patient-self
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PS128
Number analyzed (Participants) | 25
hours
  pre | 9.92 (1.76)
  psot | 10.76 (1.68)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.031, t-test, 2 sided

6. Secondary Outcome: Change in Nonmotor Symptoms: 30-item Screening Questionnaire (NMS-Quest) Total Score
Description: NMS-Quest is a 30-item Screening tool for non-motor symptoms of Parkinson's disease. The minimum total score possible is 0 and the maximum total score possible is 30. Higher values represent a worse outcome.
Time Frame: Baseline to Week 12 assessed on Medication
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PS128
Number analyzed (Participants) | 25
score on a scale
  pre | 6.84 (4.65)
  post | 6.28 (4.35)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.115, t-test, 2 sided

7. Secondary Outcome: Change in The Parkinson's Disease Questionnaire (PDQ-39)
Description: The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. The minimum possible score is 0 and the maximum possible score is 100. Higher values represent a worse outcome."
Time Frame: Baseline to Week 12 assessed on Medication
Population: Participants who completed the 12-week intervention were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PS128
Number analyzed (Participants) | 25
score on a scale
  pre | 19.86 (9.60)
  post | 14.18 (8.61)
Statistical Analysis 1: Comparison: PS128; Test type: Other; p = 0.031, t-test, 2 sided

8. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: The Patient Global Impression of Change (PGI-C) consists of one item taken from the clinical global impression and adapted to the patient. The minimum total score possible is 1 and the maximum total score possible is 7. Higher values represent a worse outcome. We exploratorily investigate participants' subjective impression after intervention by PGI-C. The percentage of participant's response in each category, such as "very much improved", "minimally improved", "no change", or "minimally worse" were used to draw an overall conclusion of the intervention potential in the open-arm trial.
Time Frame: Week 12 assessed on Medication
Population: Participants who completed the 12-week intervention were included.
Measure: Count of Participants; unit: Participants
Arm/Group | PS128
Number analyzed (Participants) | 25
Participants
  Very much improved | 1
  Much improved | 4
  Minimally improved | 12
  No change | 7
  Minimally worse | 1

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: For safety assessment, physical and neurological examinations were performed to evaluate the overall health of the subjects at weeks 0 and 12. In addition, all subjects were actively monitored for the occurrence of adverse events by telephone at least once per week.
Arm/Group | PS128
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04389762/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT04389762/ICF_002.pdf